CLINICAL TRIAL: NCT06610409
Title: Assessment of CXCL5 Level in SLE Patients and Its Correlation with Disease Activity
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Reem Amr Mohamed Essmat, Dairuit , Assuit, Assiut University
Other Study IDs: CXCL5 in SLE patients
Record Dates: First submitted 2024-09-20; First posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: SLE (Systemic Lupus)
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- SLE patients
  Interventions: Diagnostic Test: blood sampling
- Healthy controls
  Interventions: Diagnostic Test: blood sampling

INTERVENTIONS:
Diagnostic Test: blood sampling — Blood sample for CXCL5 Level

SUMMARY:
Assessment of CXCL5 biomarker in Serum of patients of SLE in comparison to healthy patients and its correlation with disease activity

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is a common autoimmune disease involving multiple organs and systems. SLE is characterized by the production of a large number of autoantibodies and the deposition of various immune complexes in target tissue .(1,2).

Chemokines are a large family of small secreted proteins that are identified as attractants of different types of leukocytes, including neutrophils, to sites of infection and inflammation. They are produced locally in tissues and act through interaction with specific G protein-coupled receptors that are predominantly expressed on leukocytes(3,4,5). Interaction between chemokines and their receptor plays an essential role in the development and homeostasis of the immune system as well as inflammatory response (6) . Although most chemokines promote locomotion of immune cells, some of them might inhibit leukocyte migration under certain circumstances (7).

We found in a study that serum CXCL5 levels were significantly lower in SLE patients than in healthy individuals and were negatively correlated with disease activity. By administering CXCL5 intravenously in a mouse model of lupus, mouse survival improved, and indices of disease activity reduced significantly(8,9). This finding suggests that homeostatic chemokines in peripheral blood might play an anti- inflammatory role and that serum levels of anti- inflammatory chemokines such as CXCL5 would be decreased in patients with autoimmune diseases (7) .

So in this study, we aim to determine level of CXCL5 in SLE patients , association of chemokine levels with demographics, clinical, and laboratory investigations of patients and its correlation with disease activity (7).

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old
* Patients who are diagnosed as SLE according to the 2012 Systemic Lupus International Collaborating Clinics (SLICC) Citeria (10,11).

Exclusion Criteria:

* age < 18 years old

  * Patients unwilling to participate in the study.
  * Patients with other autoimmune diseases.
  * Patients with malignancy or infections.
  * Pregnancy and lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 50 SLE patients and 40 healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
To assess CXCL5 level in SLE patients compared to healthy controls | 2024 -2027
To assess CXCL5 level in association with disease activity | 2024-2027

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine Assiut University, Asyut, Dairuit, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fan X, Ng CT, Guo D, Lim F, Tan JC, Law A, Goh LH, Poon ZY, Cheung A, Kong SL, Tan M, Li S, Loh A, James A, Lim T, Chen J, Thumboo J, Hwang W, Low A. Dampened Inflammation and Improved Survival After CXCL5 Administration in Murine Lupus via Myeloid and Neutrophil Pathways. Arthritis Rheumatol. 2023 Apr;75(4):553-566. doi: 10.1002/art.42383. Epub 2023 Feb 22. PMID 36240108
- [Background] Zhang L, Zhao L, Du K, Chen J, Ding H, Petersen F, Ye S, Lin Z, Yu X. Serum levels of CXCL5 are decreased and correlate with circulating platelet counts in systemic lupus erythematosus. Int J Rheum Dis. 2024 Mar;27(3):e15089. doi: 10.1111/1756-185X.15089. PMID 38439196